CLINICAL TRIAL: NCT04102514
Title: A Dyadic Approach for a Remote Physical Activity Intervention in Adults With AD and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00144595; R01AG061187 (NIH)
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Results first posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2024-08

CONDITIONS: Alzheimer Disease
Keywords: Physical Activity; Exercise
MeSH Terms: conditions — Alzheimer Disease; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real-time Group Video (Other)
  Interventions: Behavioral: Real-time Group Video
- Enhanced Usual Care (Other)
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Real-time Group Video — Dyads in the RGV arm will be asked to complete three 45 min sessions that include aerobic, resistance, and balance/coordination exercises delivered by a trained health coach via Zoom® software on an iPad during mos. 0-6, and 1 session/wk. during mos. 7-12 to groups of 5-8 dyads in their home along with being provided written materials regarding exercise and physical activity from the National Institute on Aging and brief (15-20 min) FaceTime meetings (0-6 mos.= 2/mo.; 7-12 mos.= 1/mo.) with the heath coach to discuss progress, provide support and receive additional guidance on how to increase MPA.
  Arms: Real-time Group Video
Behavioral: Enhanced Usual Care — Dyads in the EUC arm, will be given a recommended exercise plan to follow on their own along with being provided written materials regarding exercise and physical activity from the National Institute on Aging and brief (15-20 min) FaceTime meetings (0-6 mos.= 2/mo.; 7-12 mos.= 1/mo.) with the heath coach to discuss progress, provide support and receive additional guidance on how to increase MPA.
  Arms: Enhanced Usual Care

SUMMARY:
The objective of this study is to compare the effectiveness of 2 intervention delivery strategies for increasing moderate physical activity (MPA), real-time group video conferencing (RGV) vs. enhanced usual care (EUC), in community dwelling adults with Alzheimer's diseases (AD) and their caregiver (dyads) over 18 mos. (6 mos. active, 6 mos. maintenance, 6 mos. no contact). The primary outcome is to compare total MPA (min/wk.), assessed using ActiGraph, in adults with AD from baseline to 6 mos. Secondary aims for the Adults with AD are to compare MPA (min/wk), sedentary time (min/wk.), percentage meeting 150 min/wk. goal, functional fitness, activities of daily living (basic/instrumental), quality of life, residential transitions, and cognitive function across 18 months between RGV and EUC. Secondary aims for the caregivers are to compare total MPA (min/wk.), sedentary time (min/wk.), functional fitness, quality of life, caregiver burden across 18 months between RGV and EUC. Additionally, as an exploratory aim, this study will evaluate the influence of process variables/participant characteristics on MPA in adults with AD and their caregiver across 6, 12 & 18 mos.: age, sex, BMI, attendance (exercise/support sessions), use of recorded videos, PA self-monitoring, peer interactions during group sessions, caregiver support, type and quality of dyadic relationship, and number of caregivers.

DETAILED DESCRIPTION:
This study will compare 2 strategies for the delivery of an intervention to increase moderate physical activity (MPA) in community dwelling adults with AD and their caregiver (dyads); real-time group video conferencing (RGV) vs. enchanced usual care (EUC). Adults (age ≥ 55 yrs.) with mild to moderate AD (n=100) and their caregiver (n=100) will be randomized (1:1) to one of the 2 intervention arms for an 18-mo. trial (6 mos. active intervention, 6 mos. maintenance, 6 mos no contact). Cohorts of ~20 dyads will be recruited and computer randomized. Dyads will be stratified by the sex of the person with AD, and sequentially randomized by the study statistician with equal allocation to the RGV or EUC arms. Participants in both arms will be provided with an iPad® for intervention delivery, Fitbit (Fitbit Inc., San Francisco, CA) for self-monitoring MPA, and will be asked to complete 150 min of MPA/wk. Dyads in the RGV arm will be asked to complete three 45 min sessions that include aerobic, resistance, and balance/coordination exercises delivered by a trained health coach via Zoom® software on an iPad during mos. 0-6, and 1 session/wk. during mos. 7-12 to groups of 5-8 dyads in their home. Dyads in the EUC arm, will be given a recommended exercise plan to follow own their own. Dyads in both arms will be provided with written materials regarding exercise and physical activity from the National Institute on Aging and will be asked to complete brief (15-20 min) FaceTime meetings (0-6 mos.= 2/mo.; 7-12 mos.= 1/mo.) with the heath coach to discuss progress, provide support and receive additional guidance on how to increase MPA. All outcomes will be collected by trained research assistants who are blinded to the study condition. The primary outcome, total MPA, will be assessed, in both individuals with AD and caregivers, by Actigraph at baseline, 3, 6, 12 & 18 mos. All secondary/exploratory outcomes will be assessed at the individual with AD or caregivers' home at baselines, 6, 12, and 18 months. Secondary outcomes for the individual with AD are sedentary time, functional fitness, activities of daily living, quality of life, residential transition, and cognitive function. Secondary outcomes for the caregiver are sedentary time, functional fitness, quality of life, and caregiver burden. The exploratory outcomes are age, sex, BMI, attendance (exercise/support sessions), use of pre-recorded videos, PA self-monitoring, peer interactions during group sessions, caregiver support, type and quality of dyadic relationship, and number of caregivers. This trial is powered to detect a between-arm difference (RGV vs. EUC) of 10 min./d. in MPA. This difference represents additional 70 mins. of MPA/wk. in the RGV arm. Power analysis shows that 84 participants (42/arm) would provide 81% power to test an overall between-arm difference across time, i.e., group effect. This sample size would also provide ≥ 80% power to detect a between-arm difference in change, i.e., group-by-time interaction, as small as f = 0.10. Thus, conservatively assuming a high attrition rate of 20%, the study team will recruit 100 dyads at baseline to assure the final sample size requirements are achieved, i.e., final N ≥ 84 (thus, power ≥ 80%) with attrition up to 20%. General mixed modeling for repeated measures will be utilized to evaluate the primary aim to compare total MPA (min/wk.) across the 6 mo. active intervention in adults with AD and their caregiver randomized to the RGV and EUC interventions. A similar mixed modeling analysis will be conducted to examine the secondary aim. General mixed models will be fitted for the two arms combined to examine the association for the process variables/participant characteristics with MPA. However, if there is a significant between-arm difference in MPA, the investigators will determine whether the process variables/participant characteristics amplify or attenuate the RGV effect, i.e., moderation, by testing a 2-way interaction with the group effect and/or a 3-way interaction with the group-by-time interaction term.

ELIGIBILITY:
Inclusion Criteria:

Adults with AD -

1. Very mild to moderate dementia
2. Age ≥ 55 yrs
3. Low-risk of falls
4. Ability to participate in MPA, e.g., walk including with an assistive device, as verified PCP clearance.
5. Ability to communicate verbally.
6. Vision and hearing sufficient to safely comply with the intervention program as verified by PCP clearance.
7. Reside at home and receive support from a caregiver.
8. Internet access in the home.

Caregivers-

1. Age ≥18 yrs.
2. Spends at least 20 hrs./wk. with the adult with AD.

Exclusion Criteria: Adults with AD-

1. Current exercise, i.e., > 3, 30-min bouts of planned exercise/wk.
2. Clinically significant psychiatric disorder; systemic illness or infection likely to affect safety; clinically-evident stroke; myocardial infarction or coronary artery disease in the last 2 yrs.; cancer in the last 5 yrs.; or significant pain or musculoskeletal symptoms that would prohibit exercise.
3. Unwilling to be randomized.

Caregivers-

1. Unable to participate in MPA, i.e., brisk walking.
2. Unwilling to be randomized.
3. Serious medical risk, such as cancer within the last 5 yrs. or cardiac event, i.e., heart attack, stroke, angioplasty within the last 2 yrs.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2024-08-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas, Lawrence, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Real-time Group Video: Alzheimer's Patient: Alzheimer's Patients randomized to the RGV arm were asked to complete three 45 min sessions that include aerobic, resistance, and balance/coordination exercises delivered by a trained health coach via Zoom® software on an iPad during mos. 0-6, and 1 session/wk. during mos. 7-12 to groups of 5-8 dyads in their home along with being provided written materials regarding exercise and physical activity from the National Institute on Aging and brief (15-20 min) FaceTime meetings (0-6 mos.= 2/mo.; 7-12 mos.= 1/mo.) with the heath coach to discuss progress, provide support and receive additional guidance on how to increase MPA.
- Real-time Group Video: Caregiver: Caregivers of Alzheimer's patients randomized to the Real-time Group Video arm attended three 45 min sessions with the Alzheimer's Patient that included aerobic, resistance, and balance/coordination exercises delivered by a trained health coach via Zoom® software on an iPad during mos. 0-6, and 1 session/wk. during mos. 7-12 to groups of 5-8 dyads in their home along with being provided written materials regarding exercise and physical activity from the National Institute on Aging and brief (15-20 min) FaceTime meetings (0-6 mos.= 2/mo.; 7-12 mos.= 1/mo.) with the heath coach to discuss progress, provide support and receive additional guidance on how to increase MPA.
- Enhanced Usual Care: Alzheimer's Patient: Alzheimer's Patients in the EUC arm, were given a recommended exercise plan to follow on their own along with being provided written materials regarding exercise and physical activity from the National Institute on Aging and brief (15-20 min) FaceTime meetings (0-6 mos.= 2/mo.; 7-12 mos.= 1/mo.) with the heath coach to discuss progress, provide support and receive additional guidance on how to increase MPA.
- Enhanced Usual Care: Caregiver: Caregivers in the EUC arm, assisted the Alzheimer's Patient with increasing MPA and were given a recommended exercise plan to follow on their own along with being provided written materials regarding exercise and physical activity from the National Institute on Aging and brief (15-20 min) FaceTime meetings (0-6 mos.= 2/mo.; 7-12 mos.= 1/mo.) with the heath coach to discuss progress, provide support and receive additional guidance on how to increase MPA.
Period: Overall Study
Arm/Group | Real-time Group Video: Alzheimer's Patient | Real-time Group Video: Caregiver | Enhanced Usual Care: Alzheimer's Patient | Enhanced Usual Care: Caregiver
Started | 57 | 57 | 42 | 42
Completed | 41 | 44 | 27 | 28
Not Completed | 16 | 13 | 15 | 14
Not completed — Death | 3 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 3 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 7 | 13 | 7 | 14
Not completed — Moved to longterm care facility | 6 | 0 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Real-time Group Video: Alzheimer's Patient | Real-time Group Video: Caregiver | Enhanced Usual Care: Alzheimer's Patient | Enhanced Usual Care: Caregiver | Total
Number analyzed (Participants) | 57 | 57 | 42 | 42 | 198
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 16 | 4 | 9 | 38
  >=65 years | 48 | 41 | 38 | 33 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.0 (8.0) | 68.5 (11.8) | 75.8 (8.6) | 69.7 (12.1) | 73.5 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 38 | 16 | 31 | 108
  Male | 34 | 19 | 26 | 11 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 3 | 4 | 9
  Not Hispanic or Latino | 56 | 56 | 39 | 38 | 189
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 1 | 7
  White | 53 | 53 | 40 | 40 | 186
  More than one race | 1 | 1 | 0 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 57 | 57 | 42 | 42 | 198

OUTCOME MEASURES:

1. Primary Outcome: Moderate Physical Activity
Description: Moderate physical activity will be assessed using an ActiGraph model wGT3x-BT triaxial at baseline, 3, 6, 12 and 18 months. The ActiGraph wGT3x-BT is worn on a belt on the non-dominant hip during all waking hours for one week (7 consecutive days), with the exception of bathing, and swimming. The device measures acceleration. The acceleration values are used to determine levels of physical activity using previously validated cutpoints. Data were considered valid if they wore the accelerometer for at least 8 hours on 3 days, including 1 weekend day.
Time Frame: Baseline to 18 months
Population: Overall number of participants differs from Number analyzed below due to patients and caregivers not meeting wear-time criteria for valid data. Only those with valid wear-time were included in analysis. Additionally, participant/caregiver withdrawal resulted in differing numbers.
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Real-time Group Video: Alzheimer's Patient | Real-time Group Video: Caregiver | Enhanced Usual Care: Alzheimer's Patient | Enhanced Usual Care: Caregiver
Number analyzed (Participants) | 57 | 57 | 42 | 42
minutes per day
  Baseline Moderate Physical Activity: number analyzed (Participants) | 47 | 53 | 34 | 37
  Baseline Moderate Physical Activity | 13.3 (13.2) | 20.7 (17.5) | 14.4 (17.3) | 19.3 (19.5)
  Month 3 Moderate Physical Activity: number analyzed (Participants) | 43 | 48 | 29 | 31
  Month 3 Moderate Physical Activity | 14.7 (16.5) | 25.1 (23.2) | 11.7 (14.2) | 23.7 (21.9)
  Month 6 Moderate Physical Activity: number analyzed (Participants) | 42 | 46 | 30 | 31
  Month 6 Moderate Physical Activity | 11.6 (12.9) | 22.6 (21.1) | 14.1 (17.7) | 21.1 (21.5)
  Month 12 Moderate Physical Activity: number analyzed (Participants) | 34 | 43 | 19 | 24
  Month 12 Moderate Physical Activity | 10.8 (15.1) | 23.6 (23.5) | 12.5 (15.1) | 19.4 (15.2)
  Month 18 Moderate Physical Activity: number analyzed (Participants) | 35 | 39 | 18 | 21
  Month 18 Moderate Physical Activity | 12.6 (18.4) | 20.9 (22.7) | 16.1 (18.5) | 29.6 (21.9)

2. Secondary Outcome: Sedentary Time
Description: Sedentary time will be assessed using an ActiGraph model wGT3x-BT triaxial at baseline, 6, 12 and 18 months.
Time Frame: Baseline to 18 months
Population: Overall number of participants differs from Number analyzed below due to patients not meeting wear-time criteria for valid data. Only those with valid wear-time were included in analysis. Additionally, participant withdrawal resulted in differing numbers. This measure is for sedentary time of patients, only. Caregiver sedentary time can be found in secondary outcome 8.
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Real-time Group Video: Alzheimer's Patient | Enhanced Usual Care: Alzheimer's Patient
Number analyzed (Participants) | 57 | 42
minutes per day
  Baseline Sedentary Time: number analyzed (Participants) | 47 | 34
  Baseline Sedentary Time | 524.8 (143.3) | 590.1 (158.7)
  Month 3 Sedentary Time: number analyzed (Participants) | 43 | 29
  Month 3 Sedentary Time | 532.1 (150.6) | 577.2 (175.6)
  Month 6 Sedentary Time: number analyzed (Participants) | 42 | 30
  Month 6 Sedentary Time | 552.5 (129.5) | 601.4 (137.0)
  Month 12 Sedentary Time: number analyzed (Participants) | 34 | 19
  Month 12 Sedentary Time | 554.8 (122.1) | 647.3 (355.1)
  Month 18 Sedentary Time: number analyzed (Participants) | 35 | 18
  Month 18 Sedentary Time | 546.8 (108.6) | 521.9 (109.6)

3. Secondary Outcome: Functional Fitness
Description: Functional fitness will be measured at baseline, 6, 12 and 18 months using Functional Fitness Test (FFT) previously called the Senior Fitness Test. The individual fitness test items involve common activities such as getting up from a chair, walking, lifting, bending, and stretching.
Time Frame: Baseline to 18 months
Population: Number Analyzed differs from baseline at subsequent timepoints due to participant drops and missed data collection.
Measure: Mean (Standard Deviation); unit: Repetitions
Arm/Group | Real-time Group Video: Alzheimer's Patient | Enhanced Usual Care: Alzheimer's Patient
Number analyzed (Participants) | 57 | 42
Repetitions
  Baseline Step Test | 66.8 (28.4) | 59.4 (21.9)
  6 Month Step Test: number analyzed (Participants) | 49 | 35
  6 Month Step Test | 76.9 (28.3) | 62.2 (20.3)
  12 Month Step Test: number analyzed (Participants) | 48 | 26
  12 Month Step Test | 74.9 (28.9) | 66.7 (19.5)
  18 Month Step Test: number analyzed (Participants) | 37 | 24
  18 Month Step Test | 73.3 (25.6) | 73.3 (17.5)

4. Secondary Outcome: Activities of Daily Living
Description: Activities of daily living will be assessed at baseline, 6, 12 and 18 months using the Disabilities Assessment for Dementia (DAD). The DAD includes 40 items: 17 related to basic self-care and 23 to instrumental activities of daily living. Scores range from 0-40, with higher scores indicating less disability.
Time Frame: Baseline to 18 months
Population: Number Analyzed differs from overall analyzed due to participant drops and non-returned data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Real-time Group Video: Alzheimer's Patient | Enhanced Usual Care: Alzheimer's Patient
Number analyzed (Participants) | 57 | 42
score on a scale
  Baseline Activities of Daily Living: number analyzed (Participants) | 53 | 41
  Baseline Activities of Daily Living | 34.0 (8.8) | 30.8 (12.4)
  6 Month Activities of Daily Living: number analyzed (Participants) | 40 | 27
  6 Month Activities of Daily Living | 31.3 (11.8) | 28.7 (11.6)
  12 Month Activities of Daily Living: number analyzed (Participants) | 28 | 18
  12 Month Activities of Daily Living | 28.2 (12.4) | 29.3 (10.2)
  18 Month Activities of Daily Living: number analyzed (Participants) | 16 | 13
  18 Month Activities of Daily Living | 29.0 (14.7) | 32.7 (12.8)

5. Secondary Outcome: Change in Quality of Life
Description: Quality of life will be assessed at baseline to 18 months using the QOL-AD, a brief, 13-item self-report and 15-item caregiver-report. Each item is rated on a scale from 1-4, 1=Poor, 2=Fair, 3=Good, 4=Excellent. Scores range from 13-52, with larger numbers indicating better quality of life.
Time Frame: Baseline to 18 months
Population: Number analyzed differs from overall participants due to participant drops and non-returned surveys. Measure only pertained to Alzheimer's Patient.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Real-time Group Video: Alzheimer's Patient | Enhanced Usual Care: Alzheimer's Patient
Number analyzed (Participants) | 57 | 42
Score on a scale
  Baseline Quality of Life: number analyzed (Participants) | 53 | 41
  Baseline Quality of Life | 37.59 (4.92) | 38.61 (5.03)
  6 Month Quality of Life: number analyzed (Participants) | 40 | 27
  6 Month Quality of Life | 38.83 (5.78) | 38.75 (4.29)
  12 Month Quality of Life: number analyzed (Participants) | 28 | 18
  12 Month Quality of Life | 37.93 (5.09) | 38.81 (4.94)
  18 Month Quality of Life: number analyzed (Participants) | 16 | 13
  18 Month Quality of Life | 36.71 (5.06) | 38.30 (3.82)

6. Secondary Outcome: Residential Transitions
Description: Residential transitions, i.e., from home to institutional care, will be tracked by health coaches. Caregiver desire to institutionalize the adult with AD will be assessed using the 6-item Morycz's Desire-to-Institutionalize Scale
Time Frame: Baseline to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Real-time Group Video: Alzheimer's Patient | Enhanced Usual Care: Alzheimer's Patient
Number analyzed (Participants) | 57 | 42
Participants
  6 Month Transitions | 0 | 0
  12 Month Transitions | 2 | 3
  18 Month Transitions | 5 | 3

7. Secondary Outcome: Cognitive Function
Description: Cognitive function will be assessed at baseline, 6, 12 and 18 months using Applied Cognition Abilities 4a instruments from the Patient-Reported Outcomes Measurement Information System (PROMIS) Cognitive Function Battery. Both test contain 4 questions that will be answered by the adult with AD. Scores range from 0-100, with higher scores indicating better cognitive function.
Time Frame: Baseline to 18 months
Population: Number analyzed below differs from overall due to participant drops and non-returned data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Real-time Group Video: Alzheimer's Patient | Enhanced Usual Care: Alzheimer's Patient
Number analyzed (Participants) | 57 | 42
score on a scale
  Baseline Cognitive Function: number analyzed (Participants) | 53 | 41
  Baseline Cognitive Function | 38.6 (13.9) | 41.9 (10.1)
  6 Month Cognitive Function: number analyzed (Participants) | 40 | 27
  6 Month Cognitive Function | 27.3 (19.1) | 34.7 (16.8)
  12 Month Cognitive Function: number analyzed (Participants) | 28 | 18
  12 Month Cognitive Function | 31.8 (22.2) | 34.9 (18.5)
  18 Month Cognitive Function: number analyzed (Participants) | 16 | 13
  18 Month Cognitive Function | 24.8 (21.9) | 32.2 (19.2)

8. Secondary Outcome: Caregiver Sedentary Time
Description: Caregiver sedentary time will be assessed using an ActiGraph model wGT3x-BT triaxial at baseline, 6, 12 and 18 months.
Time Frame: Baseline to 18 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Real-time Group Video: Caregiver | Enhanced Usual Care: Caregiver
Number analyzed (Participants) | 57 | 42
minutes per day
  Baseline Sedentary Time: number analyzed (Participants) | 53 | 37
  Baseline Sedentary Time | 525.1 (143.7) | 526.9 (123.7)
  6 Month Sedentary Time: number analyzed (Participants) | 48 | 31
  6 Month Sedentary Time | 518.7 (131.4) | 526.0 (141.2)
  12 Month Sedentary Time: number analyzed (Participants) | 46 | 31
  12 Month Sedentary Time | 521.2 (116.9) | 542.1 (138.9)
  18 Month Sedentary Time: number analyzed (Participants) | 43 | 24
  18 Month Sedentary Time | 517.9 (109.6) | 571.2 (386.7)

9. Secondary Outcome: Caregiver Functional Fitness
Description: Caregiver functional fitness will be measured at baseline, 6, 12 and 18 months using Functional Fitness Test (FFT) previously called the Senior Fitness Test. The individual fitness test items involve common activities such as getting up from a chair, walking, lifting, bending, and stretching.
Time Frame: Baseline to 18 months
Population: Number Analyzed differs from baseline at subsequent timepoints due to participant drops and missed data collection.
Measure: Mean (Standard Deviation); unit: Reptetitions
Arm/Group | Real-time Group Video: Caregiver | Enhanced Usual Care: Caregiver
Number analyzed (Participants) | 57 | 42
Reptetitions
  Baseline Step Test | 80.2 (22.0) | 80.0 (20.5)
  6 Month Step Test: number analyzed (Participants) | 48 | 35
  6 Month Step Test | 94.7 (25.8) | 84.3 (19.4)
  12 Month Step Test: number analyzed (Participants) | 49 | 27
  12 Month Step Test | 93.9 (28.7) | 87.1 (20.3)
  18 Month Step Test: number analyzed (Participants) | 37 | 24
  18 Month Step Test | 96.4 (25.7) | 92.4 (22.1)

10. Secondary Outcome: Caregiver Quality of Life
Description: Caregiver quality of life will be assessed at baseline, 6, 12 and 18 months using the SF-36, which involves 36 questions relating to quality of life in typically developed adults. Scores range from 0-100, with higher score indicates better health.
Time Frame: Baseline to 18 months
Population: Number analyzed below differs from overall number due to participant drops and non-returned data. Measure only collected from Caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Real-time Group Video: Caregiver | Enhanced Usual Care: Caregiver
Number analyzed (Participants) | 57 | 42
score on a scale
  Baseline Caregiver Quality of Life: number analyzed (Participants) | 50 | 35
  Baseline Caregiver Quality of Life | 36.4 (5.8) | 37.0 (7.4)
  6 Month Caregiver Quality of Life: number analyzed (Participants) | 37 | 24
  6 Month Caregiver Quality of Life | 36.4 (7.1) | 36.3 (6.0)
  12 Month Caregiver Quality of Life: number analyzed (Participants) | 33 | 18
  12 Month Caregiver Quality of Life | 36.6 (6.5) | 37.9 (6.8)
  18 Month Caregiver Quality of Life: number analyzed (Participants) | 30 | 18
  18 Month Caregiver Quality of Life | 34.1 (6.0) | 38.1 (7.7)

11. Secondary Outcome: Caregiver Burden
Description: Caregiver Burden will be assessed at baseline, 6, 12 and 18 months using the Zarit Burden Interview-short version, a 12-item self-report questionnaire in which the caregiver is asked to answer using a 5-point scale. Scores range from 0-48, with lower scores indicating less caregiver burden.
Time Frame: Baseline to 18 months
Population: Number analyzed differs from overall due to participant drops and non-returned data. Measure was collected from Caregivers only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Real-time Group Video: Caregiver | Enhanced Usual Care: Caregiver
Number analyzed (Participants) | 57 | 42
score on a scale
  Baseline Caregiver Burden: number analyzed (Participants) | 57 | 41
  Baseline Caregiver Burden | 1.75 (0.94) | 1.49 (1.02)
  6 Month Caregiver Burden: number analyzed (Participants) | 42 | 30
  6 Month Caregiver Burden | 1.5 (0.97) | 1.53 (0.86)
  12 Month Caregiver Burden: number analyzed (Participants) | 37 | 23
  12 Month Caregiver Burden | 1.53 (0.97) | 1.52 (0.95)
  18 Month Caregiver Burden: number analyzed (Participants) | 33 | 19
  18 Month Caregiver Burden | 1.93 (1.07) | 1.28 (1.02)

12. Other Pre Specified Outcome: Body Mass Index
Description: Weight will be measured in duplicate at baseline, 6, 12 and 18 months in light clothing on a calibrated scale (Model #PS6600, Belfour, Saukville, WI) to the nearest 0.1 kg. Standing height will be measured at baseline, 6, 12 and 18 months in duplicate with a portable stadiometer (Model #IP0955, Invicta Plastics Limited, Leicester, UK). BMI will be calculated as weight (kg)/height (m2).
Time Frame: Baseline to 18 months
Population: Number analyzed below differs from overall number due to participant drops and missed data collection.
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Real-time Group Video: Alzheimer's Patient | Real-time Group Video: Caregiver | Enhanced Usual Care: Alzheimer's Patient | Enhanced Usual Care: Caregiver
Number analyzed (Participants) | 57 | 57 | 42 | 42
kg/m2
  Baseline Body Mass Index | 26.8 (4.6) | 28.4 (6.4) | 26.9 (5.3) | 29.5 (6.0)
  6 Month Body Mass Index: number analyzed (Participants) | 49 | 48 | 35 | 35
  6 Month Body Mass Index | 26.5 (4.4) | 29.0 (6.7) | 26.7 (5.1) | 29.7 (6.3)
  12 Month Body Mass Index: number analyzed (Participants) | 48 | 49 | 26 | 27
  12 Month Body Mass Index | 26.7 (4.6) | 29.1 (6.6) | 26.3 (4.9) | 29.3 (6.3)
  18 Month Body Mass Index: number analyzed (Participants) | 37 | 37 | 24 | 24
  18 Month Body Mass Index | 26.0 (3.6) | 28.8 (7.1) | 27.1 (5.0) | 28.8 (7.1)

13. Other Pre Specified Outcome: Session Attendance
Description: Session attendance for group exercise (RGV only) and support sessions will be obtained from records maintained by the health coach, and expressed as the percent of possible sessions from 0-6 mos. and 7-12 mos. Attendance for adults with AD, enrolled caregivers, and alternative caregivers will be recorded separately.
Time Frame: Baseline to 18 months
Population: Number analyzed below differs from overall number due to participant drops. Measure only collected in Real-time Group Video arm.
Measure: Mean (Standard Deviation); unit: percent of possible sessions
Arm/Group | Real-time Group Video: Alzheimer's Patient | Real-time Group Video: Caregiver
Number analyzed (Participants) | 57 | 57
percent of possible sessions
  Baseline to 6 Months | 74.0 (31.3) | 69.5 (33.0)
  Month 7 to Month 12: number analyzed (Participants) | 50 | 51
  Month 7 to Month 12 | 75.7 (46.0) | 71.0 (48.0)

14. Other Pre Specified Outcome: Use of Recorded Videos
Description: Use of recorded videos including frequency and duration of access (RGV only) will be assessed using Dropbox® analytics.
Time Frame: Baseline to 18 months
Measure: Mean (Standard Deviation); unit: Video views per week
Arm/Group | Real-time Group Video: Alzheimer's Patient | Real-time Group Video: Caregiver
Number analyzed (Participants) | 57 | 57
Video views per week | 0.17 (0.70) | 0.17 (0.70)

15. Other Pre Specified Outcome: Self-monitoring of Physical Activity
Description: Self-monitoring of physical activity will be assessed as the percentage of days with Fitbit data over a minimum of 8 hrs., between 6 am and midnight
Time Frame: Baseline to 18 months
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Caregiver Support
Description: Caregiver support will be assessed using the percentage of group exercise sessions (RGV) and/ or individual support sessions completed by both the person with AD and their caregiver.
Time Frame: Baseline to 18 months
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Peer Interactions (RGV Only)
Description: Staff will review video recordings of a random sample of 33% of group exercise sessions to identify and classify both peer to peer, and health coach to participant interactions. Interactions will be quantified and coded as verbal/non-verbal (waving, pointing, shaking head in agreement/disagreement), and as positive, neutral or negative, relative to support.
Time Frame: Baseline to 18 months
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Quality of the Dyadic Relationship
Description: Quality of the dyadic relationship will be assessed at baseline, 6, 12, and 18 mos. using the dyadic relationship scale (DRS) which measures negative and positive dyadic interactions from the perspective of both the patient and the caregiver. Scores range from 1-6, with higher scores indicating more positive dyadic relationships.
Time Frame: Baseline to 18 months
Population: Number analyzed below differs from overall number due to participant drops and non-returned data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Real-time Group Video: Caregiver | Enhanced Usual Care: Caregiver
Number analyzed (Participants) | 57 | 42
score on a scale
  Baseline Quality of the dyadic relationship: number analyzed (Participants) | 57 | 41
  Baseline Quality of the dyadic relationship | 2.69 (0.78) | 2.92 (0.66)
  6 Month Quality of the dyadic relationship: number analyzed (Participants) | 42 | 30
  6 Month Quality of the dyadic relationship | 2.71 (0.71) | 2.90 (0.55)
  12 Month Quality of the dyadic relationship: number analyzed (Participants) | 37 | 23
  12 Month Quality of the dyadic relationship | 2.72 (0.70) | 2.83 (0.65)
  18 Month Quality of the dyadic relationship: number analyzed (Participants) | 33 | 19
  18 Month Quality of the dyadic relationship | 2.72 (0.65) | 2.72 (0.75)

19. Post Hoc Outcome: Energy Expenditure of the Remote Sessions
Description: Energy expenditure of the remote sessions will be assessed using a portable metabolic system.
Time Frame: Baseline to 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Data collected over 18 month intervention.
Description: Number of participants at Risk in all categories is combined to include both Alzheimer's Patients and Caregivers.
Arm/Group | Real-time Group Video: Alzheimer's Patient | Real-time Group Video: Caregiver | Enhanced Usual Care: Alzheimer's Patient | Enhanced Usual Care: Caregiver
All-Cause Mortality (participants affected / at risk) | 3/57 | 0/57 | 0/42 | 0/42
Serious Adverse Events (participants affected / at risk) | 9/57 | 6/57 | 7/42 | 1/42
Other Adverse Events (participants affected / at risk) | 28/57 | 23/57 | 21/42 | 6/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Real-time Group Video: Alzheimer's Patient (N=57) | Real-time Group Video: Caregiver (N=57) | Enhanced Usual Care: Alzheimer's Patient (N=42) | Enhanced Usual Care: Caregiver (N=42)
Hospitalization (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 0 — Hospitalization due to fracture or muscular pain
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 0 — Respiratory hospitalization
Hospitalization (Nervous system disorders) | 3 | 0 | 0 | 0
Hospitalization (Infections and infestations) | 1 | 2 | 2 | 0
Hospitalization (Cardiac disorders) | 2 | 0 | 0 | 0
Hospitalization (Gastrointestinal disorders) | 0 | 1 | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Real-time Group Video: Alzheimer's Patient (N=57) | Real-time Group Video: Caregiver (N=57) | Enhanced Usual Care: Alzheimer's Patient (N=42) | Enhanced Usual Care: Caregiver (N=42)
Bee sting (Infections and infestations) | 1 | 0 | 0 | 0
Fall (Musculoskeletal and connective tissue disorders) | 8 | 2 | 12 | 1
Infection (Infections and infestations) | 1 | 2 | 0 | 1
Low blood pressure (Cardiac disorders) | 1 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 2 | 1
Knee pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 2 | 3
Ankle Pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 0
Hip Pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 0
Graves Disease Diagnosis (Endocrine disorders) | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0
Eye surgery (Eye disorders) | 1 | 2 | 1 | 0
Skin Cancer removal (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Arm surgery (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0 — Outpatient
Respite care (General disorders) | 1 | 0 | 0 | 0
Choking (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chronic Kidney Disease Flare Up (Renal and urinary disorders) | 0 | 1 | 0 | 0
Stepped on broken glass (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pelvic Prolapse Surgery (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 — Outpatient

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/14/NCT04102514/Prot_SAP_000.pdf